CLINICAL TRIAL: NCT03035708
Title: Human Laboratory Study of Varenicline for Alcohol Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLAB 001
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- varenicline (Experimental): 1 mg BID (2 capsules BID)
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): 1 mg BID (2 capsules BID)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Varenicline — 1 mg BID
  Other Names: Chantix
  Arms: varenicline
Drug: Placebo oral capsule — 1 mg BID
  Arms: Placebo

SUMMARY:
This study is a double-blind, randomized, placebo-controlled, parallel group, two-site study designed to assess the effects of varenicline as compared with placebo on responses to in vivo alcohol cue exposure in the human laboratory setting.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, parallel group, two-site study designed to assess the effects of varenicline as compared with placebo on responses to in vivo alcohol cue exposure in the human laboratory setting. After signing informed consent, subjects will be screened for eligibility including medical history, physical examination, vital signs, electrocardiogram (ECG), drinking history by the timeline follow-back (TLFB) method, alcohol breathalyzer test, Clinical Institute Withdrawal Assessment for Alcohol-revised (CIWA), medication use, MINI neuropsychiatric interview, urine toxicology screen, clinical chemistry, response to cue reactivity, and Columbia Suicide Severity Rating Scale (CSSR-S). Women of child-bearting potential will have a pregnancy test. If eligible for the study, subjects will be randomized using a stratified permuted block randomization procedure in an approximate 1:1 ratio (targeting 24 subjects per group - 12 subjects per group per site) to receive either varenicline or placebo for 6 weeks. Any nicotine use versus no use (cigarettes, cigars, chewing tobacco, electronic cigarettes, etc.) in the week before randomization is the stratification variable.

Varenicline or matched placebo will be titrated over the first week of the study up the maintenance dose of 1 mg (active) or two capsules (placebo) taken orally BID for an additional 5 weeks. Subjects will be seen in the clinic at screening, at randomization and 6 other times during the study. A final follow-up telephone interview will occur during Week 9 (2 weeks after the end of study visit).

After the first two weeks and after five weeks of investigational product administration at Study Week 3 and Study Week 6, respectively, subjects will undergo a cue reactivity paradigm session (HLAB) including 4 individual visual analog scale (VAS) items assessing alcohol craving, 2 VAS items assessing emotional reactivity to picture stimuli, and 2 items assessing emotional manipulation. Immediately after the HLAB session, subjects will view each picture again and record the emotion felt using the Self-Manikin Assessment (SAM).

ELIGIBILITY:
Inclusion Criteria:

To be eligible, the subject must:

* Be at least 21 years of age.
* Meet the DSM 5 criteria for alcohol use disorder of a least moderate severity (AUD-MS).
* Be seeking treatment for AUD and desire a reduction or cessation of drinking.
* Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
* Agree (if the subject is female and of child bearing potential) to use at least one of the following methods of birth control, unless she is surgically sterile, partner is surgically sterile or she is postmenopausal:

  1. oral contraceptives,
  2. contraceptive sponge,
  3. patch,
  4. double barrier (diaphragm/spermicidal or condom/spermicidal),
  5. intrauterine contraceptive system,
  6. levonorgestrel implant,
  7. medroxyprogesterone acetate contraceptive injection,
  8. complete abstinence from sexual intercourse, and/or
  9. hormonal vaginal contraceptive ring.
* Be able to take oral medication and be willing to adhere to the medication regimen.
* Complete all assessments required at screening and baseline.
* Have a place to live in the 2 weeks prior to randomization and not be at risk that s/he will lose his/her housing in the next 2 months.
* Not anticipate any significant problems with transportation arrangements or available time to travel to the study site over the next 2 months.
* Not have any unresolved legal problems that could jeopardize continuation or completion of the study.
* And others.

Exclusion Criteria:

* Contact site for additional information

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Litten, PhD, Study Director — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 23 | 24
Completed | 19 | 13
Not Completed | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.0) | 43.1 (12.1) | 43.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 15 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White | 16 | 19 | 35
  Race/ethnicity: Black | 6 | 2 | 8
  Race/ethnicity: Hispanic | 1 | 2 | 3
  Race/ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47
Drinks per day [Mean (Standard Deviation); unit: drinks/day] — Drinks per day is computed by summing the number of standard drinks consumed during the period of interest divided by the number of days in the period of interest.
  drinks/day | 6.9 (2.4) | 7.6 (2.7) | 7.3 (2.6)
Drinking per drinking day [Mean (Standard Deviation); unit: drinks/drinking day] — Drinks per drinking day is computed by summing the number of standard drinks consumed during the period of interest divided by the number of drinking days in the period of interest (i.e., days where the subject drank >0 drinks). This measure differs from the measure, drinks per day, only in the denominator (drinks per day includes all days in the period of interest).
  drinks/drinking day | 8.5 (4.1) | 9.3 (5.2) | 8.9 (4.7)
Percent days abstinent [Mean (Standard Deviation); unit: percent days abstinent] | 15.1 (16.9) | 11.8 (15.9) | 13.4 (16.3)
Percent heavy drinking days [Mean (Standard Deviation); unit: percent heavy drinking days] | 66.3 (26.5) | 71.9 (24.3) | 69.2 (25.3)
Penn Alcohol Craving Scale (PACS) score [Mean (Standard Deviation); unit: units on a scale] — The PACS is a five-item self-administered instrument for assessing alcohol craving (Flannery et al-1999). Frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking. Each item is a Likert scale ranging from 0 to 6. The items are summed to produce a total score ranging from 0 to 30. Higher total scores are indicative of greater craving.
  units on a scale | 18.0 (4.5) | 17.7 (3.8) | 17.8 (4.1)
Current smoker (past week) [Count of Participants; unit: Participants] | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cue-elicited Craving
Description: The primary outcome is cue-elicited alcohol craving, operationalized as the difference in Visual Analog Scale (VAS) craving for alcohol when exposed to an alcohol cue minus the VAS craving for alcohol when exposed to a water cue. The VAS has a minimum value of 0 and maximum value of 20; higher scores indicate more craving (a worse outcome).
Time Frame: Study Week 3
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale | 2.1 (0.4) | 2.2 (0.4)

2. Secondary Outcome: Percent Heavy Drinking Days
Description: The percentage of heavy drinking days during the last month of treatment (weeks 3-6). A heavy drinking day is defined as 4 or more drinks on a single day for females and 5 or more drinks on a single day for males.
Time Frame: Weeks 3-6
Population: mITT
Measure: Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 22 | 23
percentage of heavy drinking days | 30.7 (4.9) | 21.0 (5.0)

3. Secondary Outcome: The Percentage of Subjects Abstinent During the Last Month of Treatment (Weeks 3-6).
Description: The percentage of subjects abstinent from alcohol during the last month of treatment (weeks 3-6).
Time Frame: Weeks 3-6
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 22 | 23
Participants | 2 | 4

4. Secondary Outcome: Cigarettes Smoked Per Week
Description: The number of cigarettes smoked per week during the last month of treatment (weeks 3-6) computed only among participants who were smokers at baseline (varenicline n=11; placebo n=11). Note: cigarettes smoked per week outcome data was missing for two of the varenicline participants resulting in n=9 available for analysis.
Time Frame: Weeks 3-6
Population: mITT
Measure: Mean (Standard Error); unit: cigarettes per week
Groups:
- Varenicline - Smokers at Baseline: Subjects randomized to varenicline who smoked at baseline
- Placebo - Smokers at Baseline: Subjects randomized to placebo who smoked at baseline
Arm/Group | Varenicline - Smokers at Baseline | Placebo - Smokers at Baseline
Number analyzed (Participants) | 9 | 11
cigarettes per week | 47.0 (7.7) | 64.0 (7.6)

5. Secondary Outcome: Penn Alcohol Craving Scale
Description: Penn Alcohol Craving Scale (higher numbers are indicative of more craving for alcohol); min = 0, max = 30. The measure was assessed at Study Weeks 3, 4, 5, and 6. The reported outcome is the adjusted mean total score across weeks 3-6.
Time Frame: Study Weeks 3, 4, 5, 6 (assessed weekly during this period)
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 22 | 23
units on a scale | 10.8 (1.1) | 10.9 (1.1)

ADVERSE EVENTS:
Time Frame: Weeks 1 to 6
Description: Definitions and descriptions are consistent with those in clinicaltrials.gov.
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/24
Other Adverse Events (participants affected / at risk) | 19/23 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=23) | Placebo (N=24)
Seizure (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=23) | Placebo (N=24)
Nausea (Gastrointestinal disorders) | 10 | 4
Abnormal Dreams (Psychiatric disorders) | 7 | 5
Nasopharyngitis (General disorders) | 1 | 6
Bright Urine (Renal and urinary disorders) | 3 | 1
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Gynecological bleeding (Reproductive system and breast disorders) | 1 | 2
Headache (General disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Blurred Vision (Eye disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT03035708/Prot_SAP_000.pdf